CLINICAL TRIAL: NCT01203423
Title: Persistent Pulmonary Hypertension of the Newborn (PPHN) Observational Study
Acronym: PPHN
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Michele C. Walsh/ Lead Principal Investigator, Case Western Reserve University
Other Study IDs: NICHD-NRN-0009; U10HD027881 (NIH); U10HD021373 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD021397 (NIH); U01HD019897 (NIH); U10HD021415 (NIH); U10HD027856 (NIH); U10HD021364 (NIH); U10HD027880 (NIH); U10HD027904 (NIH); U10HD027871 (NIH); U10HD021385 (NIH); M01RR000997 (NIH); M01RR008084 (NIH); M01RR000750 (NIH); M01RR000070 (NIH); M01RR006022 (NIH)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Persistent Fetal Circulation Syndrome; Persistent Pulmonary Hypertension of Newborn
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Prematurity; Persistent Pulmonary Hypertension of Newborn (PPHN)
MeSH Terms: conditions — Premature Birth; Persistent Fetal Circulation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study was an observational study to estimate the prevalence of Persistent pulmonary hypertension of the newborn (PPHN) among term or near-term infants with severe respiratory disease.

DETAILED DESCRIPTION:
The optimal approach to the treatment of PPHN remains controversial. In 1978, hyperventilation was advocated for the treatment of PPHN. Newer therapies such as alkali infusion have been introduced without the support of randomized trial. In addition, in 1993, large controlled trials of inhaled nitric oxide were in the planning stages. There is a lack of knowledge about how these diverse management styles impact patient outcome.

Given the large number of treatments used in neonates with PPHN, we wished to document treatment of PPHN and outcomes of those treatments. Therefore, we performed a prospective, observational study to document prevalence of PPHN, the treatments and outcomes in a large population of infants treated at the 12 centers of the National Institute of Child Health and Human Development (NICHD) Neonatal Research Network. Further, we sought to compare treatment with hyperventilation to treatment with alkali infusion.

ELIGIBILITY:
Inclusion Criteria:

* >= 34 weeks gestational age
* On mechanical ventilation and/or fraction of inspired oxygen >0.50; and
* Had documented pulmonary artery hypertension as defined by either two-dimensional echocardiographic evidence of elevated pulmonary pressure (judged by right to left or bidirectional shunt), or a preductal to postductal oxygen gradient >20 mm Hg

Exclusion Criteria:

* >7 days of age

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The infants were screened within the first 24 hours and were followed until enrollment criteria were met or until they reached 7 days of age, whichever occurred first.
Sampling Method: Probability Sample
Enrollment: 385 (Actual)
Dates: Start 1993-10; Primary Completion 1994-12 (Actual); Study Completion 1994-12 (Actual)

PRIMARY OUTCOMES:
Death | 120 days of age

CONTACTS AND LOCATIONS:
Overall Officials: Michele C. Walsh, MD MS, Study Director — Case Western Reserve University; Lu-Ann Papile, MD, Principal Investigator — University of New Mexico; Jon E. Tyson, MD MPH, Principal Investigator — University of Texas; Barbara J. Stoll, MD, Principal Investigator — Emory University; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Charles R. Bauer, MD, Principal Investigator — University of Miami; Raymond Bain, PhD, Principal Investigator — George Washington University; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee at Memphis; James A. Lemons, MD, Principal Investigator — Indiana University; David K. Stevenson, MD, Principal Investigator — Stanford University; William Oh, MD, Principal Investigator — Brown University, Womens and Infants Hospital; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; Seetha Shankaran, MD, Principal Investigator — Wayne University
Locations (13):
- United States (13):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Result] Walsh-Sukys MC, Tyson JE, Wright LL, Bauer CR, Korones SB, Stevenson DK, Verter J, Stoll BJ, Lemons JA, Papile LA, Shankaran S, Donovan EF, Oh W, Ehrenkranz RA, Fanaroff AA. Persistent pulmonary hypertension of the newborn in the era before nitric oxide: practice variation and outcomes. Pediatrics. 2000 Jan;105(1 Pt 1):14-20. doi: 10.1542/peds.105.1.14. PMID 10617698
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/